CLINICAL TRIAL: NCT06704048
Title: Healthrelated Quality of Life and Experiences of a Heart Rehabilitation Programme After Care for Infective Endocarditis. a Quantitave and Qualitative Study with Mixed Methods.
Brief Title: Healthrelated Quality of Life and Experiences of a Heart Rehabilitation Programme After Care for Infective Endocarditis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Halland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-03596-01 v
Record Dates: First submitted 2024-11-14; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Infective Endocarditis; Bacterial Infections; Cardiac Rehabilitation; Patient Participation
Keywords: Infective Endocarditis; Bacterial Infections; Patient Participation; Interview; Qualitative Research; Cardiac rehabilitation
MeSH Terms: conditions — Endocarditis; Bacterial Infections; Patient Participation | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Intervention Model Description: Mixed method
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cardiac rehabilitation (Experimental): An intervention with physical exercise training within cardiac rehabilitation according to the SEPHIA and SWEDEHEART protocols is offered to a new group of patients, patients with infective endocarditis.
  The intervention is studied with qualitative and quantitative methods on regard of the physical and health-related effects of rehabilitation, the adherence to the intervention and the health restoration in general. Patient's perspectives on rehabilitation and health restoration are given in interviews.
  Interventions: Other: Cardiac rehabilitation

INTERVENTIONS:
Other: Cardiac rehabilitation — Standard hospital-based cardiac rehabilitation according to SEPHIA and SWEDEHEART protocols 2 times a week for 12 weeks with individualized physical evaluation before and after the intervention.

SUMMARY:
Can the health of patients with Infective endocarditis (IE) be improved by participation in the physical exercise training within cardiac rehabilitation program?

Participants will:

* Be physically evaluated by a physiotherapist before and after the progam of physical exercise training within cardiac rehabilitation.
* Do individual exercises in a group led by a physiotherapist 2 times weekly during 12 weeks.
* Answer digitally surveys on the perceived health for 4 times during 1 year
* Participate in interviews on patient's experiences of health and rehabilitation 1 time before and 2 times after the training program during I year.

DETAILED DESCRIPTION:
Infective endocarditis (IE) is a rare but severe infectious disease of the heart. Patients with IE are treated for weeks in the hospital and have profound impairments of health for a long time after the treatment. Patients experience a delayed recovery after discharge both physically, with wasting and fatigue; and mentally, with anxiety and depression. Patients suffer from a diminished quality of life and have difficulties returning to work, up to a year post-discharge. Little is known about how patients perceive the IE disease after discharge and if patient's health can be promoted by rehabilitation since no studies have been able to evaluate the effect of interventions aimed at relieving these problems.

The hypothesis is that physical exercise training within cardiac rehabilitation can improve physical capacity and reduce symptoms of fatigue. Other aspects of quality of life, mental health, self-rated health and the impact on anxiety and depression will also be studied.

The investigators aim to study the intervention of physical exercise training within cardiac rehabilitation on the group of patients with IE. The patients with IE will be offered physical exercise training within cardiac rehabilitation according to the protocols of SEPHIA (Secondary Prevention after Heart Intensive Care Admission), as documented in SWEDEHEART(Swedish Web-system for Enhancement and Development of Evidence-based care in Heart disease Evaluated According to Recommended Therapies).

Individualized center-based evaluations according to the protocols are performed before and after the rehabilitation period. Exercises and training are performed in groups led by specialized physiotherapists 2 times per week for 12 weeks. Surveys on health-related quality of life, symptoms of fatigue, anxiety, depression, and occupational balance are digitally distributed at 4 occasions during 1 year after IE. Qualitative interviews will be used 3 times the first year to evaluate the effect and meaning of the program on health and well-being.

Both the patients' physical improvements for 1 year after IE ( by physiotherapeutic testing) as well as the self-reported experiences of symptoms of fatigue and other aspects of health-related quality of life by surveys will be studied. The patients are also interviewed on expectations and experiences of the intervention and what the patients think is the optimal strategy to regain health. A mixed methods design is chosen to include both quantitative and qualitative data to evaluate the intervention.

50 patients treated for IE will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of infective endocarditis (IE) based on Dukes ISCVID criteria and discharged after treatment for IE from the Department of Infectious Diseases, Hospital of Halmstad, Region Halland, Sweden.

Exclusion Criteria:

* Not able to do a bicycle ergometer test or training.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2035-08 (Estimated)

PRIMARY OUTCOMES:
Quantitative - 1. Changes from test 1 before start of physical exercise training within cardiac rehabilitation to test 2 at the end of the physical exercise training period and test 3 6-12 months after the end of the physical exercise training period. | 18 months
  1 Test of maximal workload (in Watt) and time (in minutes and seconds). Submaximal exercise capacity on a symptom-limited bicycle ergometer test with an increased workload of 25W every 4.5 minutes. The exercise test is discontinued at Borg rating of perceived exertion (RPE) scale 17 and/or dyspnea 7 at Borg´s CR-10 scale.
  Pre-exercise screening test is compared to the post-exercise tests.
Quantitative - 2. Changes from test 1 before start of physical exercise training within cardiac rehabilitation to test 2 at the end of the physical exercise training period and test 3 6-12 months after the end of the physical exercise training period. | 18 months
  2 Muscular endurance tests with a unilateral isotonic shoulder flexion and a unilateral isotonic heel lift(maximum number of repetitions).
  Pre-exercise screening test is compared to the post-exercise tests.
Quantitative - 3. Changes from test 1 before start of physical exercise training within cardiac rehabilitation to test 2 at the end of the physical exercise training period and test 3 6-12 months after the end of the physical exercise training period. | 18 months
  3 Changes in symptoms of fatigue assessed by the questionnaire Mental Fatigue Inventory (MFI-20) survey.
  The MFI is a self-report instrument designed to measure symptoms of fatigue which consists of 20 items and, by which 5 dimensions can be calculated (General Fatigue (GF), Physical Fatigue (PF), Reduced Motivation (RM), Reduced Activity (RA) and Mental Fatigue (MF)).
  Pre-exercise screening test is compared to the post-exercise tests.
Quantitative - Degree of patient adherence to the program | 16 weeks
  Number of times in physical exercise-training within cardiac rehabilitation. Full adherence is set to 12 times during 16 weeks
Qualitative - Patients's experiences on cardiac rehabilitation | 0, 3 months, 6-12 months
  Qualitative content analysis of interviews before start of physical exercise training within cardiac rehabilitation, at the end of the physical exercise training period and 6-12 months after the end of the physical exercise training period.
  Descriptive.
Qualitative - Patients's experiences on post-infection health restoration | 6-12 months
  Qualitative content analysis of interviews 6-12 months after the end of the physical exercise training period.
  Descriptive.
Mixed method - Hindrances and possibilities for patients in participating after IE in physical exercise training within cardiac rehabilitation program | 12 months
  Qualitative interviews will be compared with quantitative data of participation and test result to describe and explain the findings.
Mixed method - Description and explanation on the health evolution the first year after IE among patients offered physical exercise training within cardiac rehabilitation program | 12 months
  Qualitative interviews will be compared with quantitative data of test results on physical capacity and health-related quality of life to describe and explain the findings.

OTHER OUTCOMES:
Quantitative - HADS (Hospital Anxiety and Depression Scale) as a screening tool for mental malaise | 1 year
  Evaluation and interpretation of HADS as a screening tool to find patients that benefit from intervention physically or mentally.
Quantitative - OBQ-11 (Occupational Balance Questionnaire) as a screening tool for fatigue | 1 year
  Evaluation and interpretation of OBQ-11 as a screening tool to find patients that benefit from intervention physically or mentally.
Quantitative - MFI-20 (Multidimensional Fatigue Inventory) as a screening tool for fatigue | 1 year
  Evaluation and interpretation of MFI-20 as a screening tool to find patients that benefit from intervention physically or mentally.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Larsson, PhD,Prof, Study Director — Department of Health and Nursing, School of Health and Welfare, Halmstad, Sweden; Magnus Rasmussen, MD,PhD,Prof, Study Director — Department of Clinical Sciences Lund, Division of Infection Medicine, Lund University, Lund, Sweden
Locations (1):
- Helena Lindberg, Halmstad, Halland County, Sweden

IPD SHARING:
Plan to Share IPD: No
Quantitative data can be pseudonymized and shared with other researchers upon request.

REFERENCES:
- [Background] Rasmussen TB, Zwisler AD, Risom SS, Sibilitz KL, Christensen J, Bundgaard H, Moons P, Thygesen LC, Lindschou J, Norekval TM, Berg SK. Comprehensive cardiac rehabilitation for patients following infective endocarditis: results of the randomized CopenHeartIE trial. Eur J Cardiovasc Nurs. 2022 Apr 9;21(3):261-270. doi: 10.1093/eurjcn/zvab047. PMID 34089600
- [Background] Abraham LN, Sibilitz KL, Berg SK, Tang LH, Risom SS, Lindschou J, Taylor RS, Borregaard B, Zwisler AD. Exercise-based cardiac rehabilitation for adults after heart valve surgery. Cochrane Database Syst Rev. 2021 May 7;5(5):CD010876. doi: 10.1002/14651858.CD010876.pub3. PMID 33962483
- [Background] Long L, Mordi IR, Bridges C, Sagar VA, Davies EJ, Coats AJ, Dalal H, Rees K, Singh SJ, Taylor RS. Exercise-based cardiac rehabilitation for adults with heart failure. Cochrane Database Syst Rev. 2019 Jan 29;1(1):CD003331. doi: 10.1002/14651858.CD003331.pub5. PMID 30695817
- [Background] Ogmundsdottir Michelsen H, Sjolin I, Schlyter M, Hagstrom E, Kiessling A, Henriksson P, Held C, Hag E, Nilsson L, Back M, Schiopu A, Zaman MJ, Leosdottir M. Cardiac rehabilitation after acute myocardial infarction in Sweden - evaluation of programme characteristics and adherence to European guidelines: The Perfect Cardiac Rehabilitation (Perfect-CR) study. Eur J Prev Cardiol. 2020 Jan;27(1):18-27. doi: 10.1177/2047487319865729. Epub 2019 Jul 26. PMID 31349776